CLINICAL TRIAL: NCT03134976
Title: Wound Complications in Head and Neck Surgery
Status: Completed | Type: Observational
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Matthew E. Spector, Assistant Professor of Otolaryngology- Head and Neck Surgery, University of Michigan
Other Study IDs: HUM00124347
Record Dates: First submitted 2017-04-20; First posted 2017-05-01 (Actual); Last update posted 2020-06-01 (Actual); Status verified 2020-05

CONDITIONS: Hypothyroidism; Surgery; Head and Neck Cancer; Wound Heal; Laryngeal Cancer; Laryngeal Fistula
Keywords: Salvage surgery; Head and neck cancer; Wound healing; Hypothyroidism; Levothyroxine
MeSH Terms: conditions — Hypothyroidism; Head and Neck Neoplasms; Laryngeal Neoplasms | interventions — Thyroxine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Salvage Larynx: The first group includes subjects with cancer of the voice box (laryngeal squamous cell carcinoma) that has already been treated by either chemotherapy or radiation. This group will be treated using the standard of care, which includes starting thyroid hormone replacement therapy (levothyroxine) after surgery.
  Interventions: Drug: Levothyroxine
- Non-Salvage Larynx: The second group of subjects will consist of patients who have head and neck cancer of sites other than the voice box (larynx) without prior exposure to radiation or chemotherapy who are undergoing flap reconstruction surgery. This group will not be treated with levothyroxine so long as the subject has normal thyroid function. If a subject is hypothyroid, then thyroid hormone replacement will be given as a part of routine clinical care.

INTERVENTIONS:
Drug: Levothyroxine — Immediately post-operatively, all patients undergoing laryngectomy will be started on established weight-based dosing of levothyroxine administered intravenously due to the variable enteral absorption in post-operative patients including those on continuous tube feed regimens. Standard enteral dose is 1.6 mcg/kg/day. Eighty percent of this dose (1.3 mcg/kg/day) will be given IV to account for the increased bioavailability of IV levothyroxine compared to enteral levothyroxine. The maximum dose will be 200 mcg/day. Patients previously on levothyroxine at doses lower than the above dose will changed to the aforementioned standard dose. Patients on higher doses of levothyroxine pre-operatively will be maintained on on their current dosing.
  Other Names: Synthroid; Tirosint; Levoxyl; Levothroid; Unithroid; Novothyrox
  Groups: Salvage Larynx

SUMMARY:
This is a prospective observational study evaluating wound complications following head and neck surgery. Patients undergoing major head and neck surgery will be included in the study. Patients meeting eligibility criteria will be identified by members of the University of Michigan Head and Neck Oncology Division of the Department of Otolaryngology. The primary aim of this study is to identify risk factors for poor wound healing as well as biologic markers associated with wound related complications in head and neck surgery. Most specifically, this study evaluates the effects of thyroid hormone on wound healing. This study will also evaluate pre-operative labs and comorbidities as well as reconstructive factors, post-operative labs, and other variables associated with wound healing. All interventions regarding wound healing fall under current standards of care and standard practice. Data regarding post-operative wound complications will be collected in a prospective fashion on the variables under study using study-specific datasheets. Data sheet will be entered into a secure database for analysis.

ELIGIBILITY:
Inclusion Criteria:

* In both groups: subjects must be 18 years or older with biopsy confirmed cancer of the head and neck.

Exclusion Criteria:

* Children and vulnerable populations are not eligible for participation. Patients undergoing functional (non cancer related) surgery, patients who have undergone more than 1 course of radiation to the head and neck, patients with a history of thyroid cancer, patients presenting initially with a malignant fistula, patients with previous intolerance or allergy to levothyroxine, and patients without a cancer diagnosis are not eligible. Patients may enroll if they are currently hypothyroid, but will be excluded from the study if thyroid function is not normalized by the time of surgery.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients presenting to the University of Michigan Department of Otolaryngology- Head and Neck Surgery.
Sampling Method: Non-Probability Sample
Enrollment: 51 (Actual)
Dates: Start 2017-05-01 (Actual); Primary Completion 2020-04-01 (Actual); Study Completion 2020-05-01 (Actual)

PRIMARY OUTCOMES:
Number of patients treated with Levothyroxine who develop pharyngocutaneous fistula after salvage laryngectomy | 30 days post-operatively
  Blood will be drawn and analyzed for thyroid stimulating hormone (TSH), free T3, and free T4 levels at specified intervals. Subjects will be monitored for pharyngocutaneous fistula formation.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No